CLINICAL TRIAL: NCT02360111
Title: A Pilot Trial of GVHD Prophylaxis With Post Transplant Cyclophosphamide for Patients With Renal Insufficiency Undergoing a Conventional 8/8 HLA-matched Related or Unrelated Donor Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: GVHD Prophylaxis With Post Transplant Cyclophosphamide for Patients With Renal Insufficiency Undergoing a Conventional 8/8 HLA-matched Related or Unrelated Donor Allogeneic Hematopoietic Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-273
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
Keywords: GVHD Prophylaxis; Cyclophosphamide; Renal Insufficiency; Hematopoietic Stem Cell Transplant; 14-273
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Renal Insufficiency | interventions — Cyclophosphamide

ARMS (1):
- Post Transplant Cyclophosphamide (Experimental): Melphalan 70 mg/m 2/d will be administered intravenously on d-6 and -5 Fludarabine 25 mg/m 2/d will be administered intravenously on d-6 thru -2 Day -1 will be a day or rest Cyclophosphamide and mesna will be given on d+3 and +4 Siro +/- MMF will be started in those patients who are to receive it on d+5. Neupogen will begin d+7.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide

SUMMARY:
This is a pilot study which will be done in a small number of patients. The purpose of this study is to test the safety and benefit of giving a type of chemotherapy - cyclophosphamide - after the transplant to prevent graft versus host disease (GVHD) in patients with abnormal kidney function. GVHD is one of the most common complications of a stem cell transplant .

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients over age 18 who are deemed eligible for transplant by their treating physician.
* Disease status:

  1. AML in ≥ 1st remission - excluding those in 1st remission with 'good risk' cytogenetic features (i.e. t(8;21), t(15;17), inv 16).
  2. Secondary AML
  3. ALL/LL in 1st remission with clinical or molecular features indicating a high risk for relapse; or ALL > 2nd remission
  4. CML failing to respond to, progressing on or not tolerating appropriate TKI therapy in first chronic phase of disease; CML in accelerated phase, second chronic phase, or in CR after accelerated phase or blast crisis.
  5. Non-Hodgkins lymphoma with chemoresponsive disease in any of the following categories:

     1. high grade lymphomas who have failed to achieve a first CR or have relapsed following a 1st remission who are not candidates for autologous transplants or transplants requiring the use of calcineurin inhibitors.
     2. any NHL with therapy responsive disease which is considered not curable outside the transplant setting and not eligible/appropriate for autologous transplant or a higher priority protocol.
  6. Myelodysplastic syndrome (MDS): RA/RCMD with high risk cytogenetic features or transfusion dependence, RAEB-1 and RAEB-2 and AML evolved from MDS, who are not eligible for a higher priority protocol.
  7. Chronic myelomonocytic leukemia: CMML-1 and CMML-2, advanced polycythemia vera, and myelofibrosis.

     1. Patients must have a healthy HLA compatible (8/8 molecularly matched related, or unrelated) donor willing to undergo BM harvesting or PBSC apheresis after G-CSF administration. BM will be the preferred graft source.
     2. Patients diagnosed with any form of acute leukemia must have received induction and at least one course of consolidation chemotherapy pretransplant
* Patients must have a Karnofsky Performance Status > 70%
* Patients will have a eGFR <60 ml/min/1.73 m2

  1. Patients must have adequate organ function measured by: Cardiac: asymptomatic or if symptomatic then LVEF at rest must be > 50% and must improve with exercise.
  2. Hepatic: ALT < 3 x ULN and total serum bilirubin < 1.5 x ULN, unless there is congenital benign hyperbilirubinemia
  3. Renal: eGFR > 30 ml/min/1.73 m2
  4. Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)
* Each patient must be willing to participate as a research subject and must sign an informed consent form.
* Patient must have a fully matched related or unrelated donor willing to donate stem cells.

Exclusion Criteria:

* Major surgery or irradiation within two weeks.
* Active CNS or extramedullary malignant disease.
* Active and uncontrolled infection at time of transplantation including active infection with Aspergillus or other mold, or HIV infection
* Pregnant or lactating women - they are excluded, given the potential teratogenic effects of chemotherapy and agents used in the transplant.
* Male and female patients of child-bearing potential unwilling to use effective means of contraception
* HIV or HTLV I/II positive, hepatitis C or chronic active hepatitis B.
* Patients who have had a previous malignancy unless they are deemed by their treating physicians to be at low risk for recurrence.
* Patient or guardian unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up and research tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Jakubowski, Ph.D., M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Post Transplant Cyclophosphamide: Melphalan 70 mg/m 2/d will be administered intravenously on d-6 and -5 Fludarabine 25 mg/m 2/d will be administered intravenously on d-6 thru -2 Day -1 will be a day or rest Cyclophosphamide and mesna will be given on d+3 and +4 Siro +/- MMF will be started in those patients who are to receive it on d+5. Neupogen will begin d+7.
  Cyclophosphamide
Period: Overall Study
Arm/Group | Post Transplant Cyclophosphamide
Started | 3
Completed | 1
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Post Transplant Cyclophosphamide
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 70 [64 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: # GVHD (Grade II-IV) Chronic GVHD Will be Diagnosed and Graded According to the (NIH Criteria)
Description: Chronic GVHD will be diagnosed and graded according to the (NIH criteria) treated with standard or experimental immunosuppressive therapy.
Time Frame: 2 years
Population: Protocol terminated prematurely due to low accrual
Arm/Group | Post Transplant Cyclophosphamide
Number analyzed (Participants) | 0

2. Secondary Outcome: Disease-free Survival
Description: DFS is defined as the minimum interval of time to relapse/recurrence, to death or to the last follow-up, from the time of transplant
Time Frame: 2 years
Population: Protocol terminated prematurely due to low accrual
Arm/Group | Post Transplant Cyclophosphamide
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from transplant to death or last follow-up.
Time Frame: 2 years
Population: Protocol terminated prematurely due to low accrual
Arm/Group | Post Transplant Cyclophosphamide
Number analyzed (Participants) | 0

4. Secondary Outcome: # Renal Insufficiency Defined as a Calculated eGFR <60 ml/Min/1.73m2. Those With a eGFR < 30 ml/Min/1.73m2 Will be Considered Ineligible.
Description: Renal insufficiency is defined as a calculated eGFR <60 ml/min/1.73m2. Those with a eGFR < 30 ml/min/1.73m2 will be considered ineligible.
Time Frame: 2 years
Population: Protocol terminated prematurely due to low accrual
Arm/Group | Post Transplant Cyclophosphamide
Number analyzed (Participants) | 0

5. Secondary Outcome: The Occurrence of Life-threatening Opportunistic Infections
Description: will be evaluated according to the criteria established by BMT CTN , and will be correlated with the level of immune recovery.
Time Frame: 2 years
Population: Protocol terminated prematurely due to low accrual
Arm/Group | Post Transplant Cyclophosphamide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Post Transplant Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Post Transplant Cyclophosphamide (N=3)
Acute kidney injury (Renal and urinary disorders) | 1
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 2
Pericardial effusion (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Salivary gland infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Urinary retention (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Post Transplant Cyclophosphamide (N=3)
Anemia (Blood and lymphatic system disorders) | 3
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
White blood cell decreased (Investigations) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Lung infection (Infections and infestations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT02360111/Prot_SAP_000.pdf